CLINICAL TRIAL: NCT06686732
Title: Effect Of Multimodal Approach On Rehabilitation Of The Patient With Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Multimodal Rehabilitation Approach in Patients of Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS/REC/MS-PT/01939
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Lateral Epicondylitis
Keywords: tennis elbow; manual therapy; multimodal treatment; hand strength
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal group (Experimental): Experimental group included cold pack over lateral epicondyle, Passive stretching exercises in cervical spine and upper limb. Eccentric exercise of the extensor muscles associated with mobilization with movement.Neuromusclar Rehabilitation Excersise. Inhibition of points of tension in the belly of the extensor region. Early mobilization with movement with the wrist in extension. Lateral sustained glide.
  Interventions: Other: Multimodal physiotherapy
- Conventional physiotherapy (Active Comparator): Control group included Cold pack, Extensor carpi radialis brevis stretching. Active ROM of wrist flexion and extension. Active ROM of elbow flexion, extension, supination and pronation. Manually resisting wrist extensors. Maitland elbow joint mobilization with 1 min of rest between sets.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Multimodal physiotherapy — Experimental group included cold pack over lateral epicondyle. Passive stretching exercises in trapezius and levator scapulae and upper ECRB,ECRL,ECU,Extensor Digitorum, Extensor Digiti Minimi. Eccentric exercise of the extensor muscles associated with mobilization with movement. Neuromusclar Rehabilitation Excersise. In the region of origin of the tendons of the extensor muscles of the wrist and fingers for 2 min and inhibition of points of tension in the belly of the extensor region. Early mobilization with movement with the wrist in extension. Lateral sustained glide will be give at humeroradial joint during movement.
  Arms: Multimodal group
Other: Conventional physiotherapy — Control group included Cold pack for 10 mins on the lateral epicondylitis, Extensor carpi radialis brevis stretching (hold for 15 seconds x 4 reps) Active ROM of wrist flexion and extension (10 reps x 3 sets) Active ROM of elbow flexion, extension, supination and pronation (10 reps x 3 sets) . Manually resisting wrist extensors (10 second hold x 5 reps x 3 sets) 4 sets of Maitland elbow joint mobilization with 1 min of rest between sets. Baseline Dynamometer for grip strength and VAS for pain. These pre and post intervention values were mentioned in questionnaire. The participants were administered with the protocol and data was collected again immediately after the interventions without any delay.
  Arms: Conventional physiotherapy

SUMMARY:
Literature is scarce for high quality evidence regarding multimodal rehabilitation in lateral epicondylitis. By making comparisons with the conventional treatment of patients with lateral epicondylitis, the current study aims to further establish the efficacy of the multimodal rehabilitation protocol through a RCT in order to generalize the results, using dynamometer as an additional tool for pre and post assessments against the outcome measures. Remarks A randomized control trial was conducted at Physical therapy departments of twin cities. The sample size was 40 calculated through G- power tool. The participants were divided into two interventional groups each having 20 participants. The study duration was eight months. Sampling technique applied was non- probability convience sampling. People of age 18-45 years, with localized point tenderness at lateral epicondyle with Mills, Cozen and Maudselys test positive were included in this research. Tools used in this study are Visual Analogue Scale, Dynamometer, Patient Rated Tennis Elbow Questionnaire. Data was collected before and immediately after the application of interventions. Data analyzed through SPSS version 23.

DETAILED DESCRIPTION:
Lateral epicondylitis is the most common lesion of the elbow complex. Despite also being referred to as "tennis elbow", lateral epicondylitis is present in less than 5-10 % of players and can appear in various tasks of excessive and repetitive effort involving movements gripping or pronation-supination.These specific patterned movements put manual laborers at the highest risk of developing lateral epicondylitis. Magnetic Resonance Imaging studies done to evaluate the prevalence of lateral epicondylitis suggest signal changes in the Extensor Carpi Radialis Brevis tendon consistent with lateral epicondylitis increase with age, with the incidence starting after 18 years of age and the peak prevalence in the subsequent decades of life. The cadaveric studies have established the direct contact of Extensor Carpi Radialis Brevis tendon with the elbow joint capsule, making it the epicondylar tendon bearing the greatest load in executing a backhand while playing tennis. Another study observed friction between the ECRB tendon and capitellum during flexion extension at the elbow joint. The Extensor Carpi Radialis Longus is the next most affected muscle in lateral epicondylitis since it has a tendon footprint 13 times greater than the Extensor Carpi Radialis Brevis on the epicondyle. As per the natural history of the lateral epicondylitis, it resolves spontaneously in 1-2 years without treatment. However, very few studies have compared outcomes with and without treatment. In a meta-analysis, no difference between nonoperative versus no treatment group was found for patients with lateral epicondylitis. One study reported no difference for the physiotherapy and corticosteroid groups compared to the wait-and-see group at 1 year against outcomes, while in another study the outcomes in the physiotherapy group were only slightly better. There are a number of different physiotherapy treatment options are available for lateral epicondylitis. However, literature is scarce for established efficacy of these treatments, largely due to lack of homogeneity as well as varied protocols of dosage and frequency. Nevertheless, these treatment options include but are not limited to stretching exercises, mobilization, electrotherapeutic modalities, deep transverse massage, orthoses, acupuncture, eccentric exercises and neuromuscular rehabilitation excercises etc. Neuromuscular rehabilitation can enhance grip strength by targeting both the muscles and the nervous system. It involves exercises that improve muscle coordination, motor control, and strength, which are crucial for a strong grip. Additionally, neuromuscular training can help re-establish proper firing patterns between the brain and muscles, leading to more efficient muscle recruitment and ultimately, improved grip strength. The treatment principle in most of these options is to reduce the force acting at the origin of the extensor muscles of the wrist allowing time for recovery to occur. The outcome reported as a result of the intervention is an improvement in pain, function and grip strength. As already stated, the available literature for the efficacy of conservative management of lateral epicondylitis cites lack of uniform results and therefore advocates for further research to establish the effect of these interventions. One such study by Marcolino et. al employed a multimodal rehabilitation protocol for lateral epicondylitis in a form of case series. This aim study aim at verifying "the efficiency of the multimodal treatment with mobilization with movement associated with eccentric strengthening, transverse massage and stretching in the treatment of eight volunteers with symptoms of lateral epicondylitis". According to this study, the results showed statistical differences in pain symptoms before and after treatment, in the analysis and functional assessment. However, lack of control group as well as the study design and the small sample size serve as confounding variables thereby limiting the ability of this study to generalize their findings. Furthermore, the study lacked objective evaluation for the assessment of grip strength. Therefore, the current study aims to work on the limitations of the study done by Marcolino et. al, by reducing the risk of biasness and eliminating the confounding variables. This will be done by conducting a randomized controlled trial in a larger sample size and comparing the suggested multimodal approach to the conventional protocol followed for lateral epicondylitis. Furthermore, in order to accurately measure the change in grip strength following the treatment protocol, dynamometer will be used.

ELIGIBILITY:
Inclusion Criteria:

* Point tenderness at the lateral epicondyle
* Positive Cozen test, Mill's test and Maudsely's test
* Symptoms duration of minimum 2 months
* Consenting to participate in the study

Exclusion Criteria:

* History of fracture in elbow, wrist or hand
* History of surgery in elbow, wrist or hand region
* Elbow conditions other than lateral epicondylitis
* Cognitive deficits and not giving consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | Three Weeks
  Changes from Baseline grip strength were taken with the help of dynamomter that measures grip strength.

SECONDARY OUTCOMES:
Visual Analogue Scale | Three Weeks
  Changes from the baseline pain levelesthe basis were measured through visual analogue scale.
Patient Rated Tennis Elbow Questionnaire | Three Weeks
  Changes in the functional Activities were noted through Patient Rated Tennis Elbow Questionnaire from the baseline and post treatment readings.

CONTACTS AND LOCATIONS:
Overall Officials: Ramsha Tariq, MS*, Principal Investigator — Riphah International University, Islamabad
Locations (3):
- Pakistan (3):
  - Muzaffar Khan Medical & Children Hospital, Wāh, Punjab Province
  - Riphah International Hospital, Sihala, Islamabad
  - DSK Physio & Rehab Center, Rawalpindi

IPD SHARING:
Plan to Share IPD: No